CLINICAL TRIAL: NCT02566551
Title: Prospective Controlled Randomized Study of Prostatic Arteries Embolization (PAE) vs Transurethral Resection of the Prostate (TURP) for Benign Prostatic Hyperplasia (BPH) Treatment.
Brief Title: Prospective Controlled Randomized Study of PAE vs TURP for BPH Treatment.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Group of Research in Minimally Invasive Techniques (Other)
Collaborators: Hospital Clínico Universitario Lozano Blesa (Other); Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, José A. Guirola, MD, MD, Group of Research in Minimally Invasive Techniques
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTM-02
Record Dates: First submitted 2015-08-10; First posted 2015-10-02 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostatic artery embolization; Transurethral resection of the prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate artery embolization (Experimental): Prostatic artery embolization (PAE) To perform embolization, gelatin microspheres (300-500 microns) will be used in this arm
  Interventions: Procedure: PAE; Device: Gelatin microspheres
- Transurethral resection of the prostate (Active Comparator): Transurethral resection of the prostate (TURP) A bipolar electrosurgery generator will be used to perform TURP
  Interventions: Procedure: TURP; Device: Bipolar electrosurgery generator

INTERVENTIONS:
Procedure: PAE — Embolization of the prostate with gelatin embolization spheres via microcatheterization of the prostatic arteries.
  Other Names: Prostate artery embolization; Prostate arteries embolization; Embolization of the prostate; Prostatic artery embolization
  Arms: Prostate artery embolization
Device: Gelatin microspheres — Gelatin embolization microspheres (300-500 microns) will be used as embolic material for the prostatic artery embolization (PAE) protocol
  Other Names: Embolization microspheres
  Arms: Prostate artery embolization
Procedure: TURP — Bipolar transurethral resection of the prostate
  Other Names: Transurethral resection of the prostate; Transurethral prostatic resection
  Arms: Transurethral resection of the prostate
Device: Bipolar electrosurgery generator — A bipolar electrosurgery generator will be used to perform transurethral resection of the prostate (TURP)
  Other Names: Transurethral prostatic resection
  Arms: Transurethral resection of the prostate

SUMMARY:
The purpose of this prospective randomized controlled study is to compare the improvement of symptoms from benign prostatic hyperplasia (BPH) and the improvement of QoL, in patients undergoing prostatic artery embolization (PAE) or conventional transurethral resection of the prostate (TURP).

DETAILED DESCRIPTION:
The purpose of this prospective randomized controlled study is to compare the improvement of symptoms from benign prostatic hyperplasia (BPH) as assessed by the International Prostate Symptom Score (IPSS) and the improvement of QoL assessed by QoL questionnaire in patients undergoing prostatic artery embolization (PAE) to patients of similar characteristics undergoing conventional transurethral resection of the prostate (TURP).

ELIGIBILITY:
Inclusion Criteria:

Patients evaluated in the Urology Service because of BPH, candidate to TURP.

* Signed informed consent
* Lower urinary tract symptoms (LUTS) secondary to BPH for at least 6 months prior to study AND/OR baseline IPSS Score > 13 AND/OR acute urinary retention with impossibility to remove urinary catheter AND/OR BPH symptoms refractory to medical treatment or for whom medication is contraindicated, not tolerated or refused Prostate size of at least 50 grams measured by MRI
* Patient must meet ONE of the following criteria:

  1. Baseline Prostate Specific Antigen (PSA) <4 ng/mL (no prostate biopsy required)
  2. Baseline PSA >4 ng/mL and ≤10 ng/mL AND free PSA > 15% of total PSA (no prostate biopsy required)
  3. Baseline PSA >4 ng/mL and ≤10 ng/mL AND free PSA <15% of total PSA AND a negative prostate biopsy result (minimum 12 core biopsy)
  4. Baseline PSA >10 ng/mL AND a negative prostate biopsy (minimum 12 core biopsy)

Exclusion Criteria:

* Active urinary tract infection
* Patients with cystoscopy findings suspicious for bladder cancer must undergo biopsy and have a negative histopathology report to be enrolled in the study
* Biopsy proven prostate or bladder cancer
* The following patients must undergo prostate biopsy with a minimum of 12 cores and have a negative histopathology report to be enrolled in the study:

  * Patients with digital rectal examination (DRE) findings suspicious for prostate cancer
  * Patients with baseline PSA levels > 10 ng/mL
  * Patients with baseline PSA levels >4 ng/mL and < 10 ng/mL AND free PSA < 15% of total PSA
* Bladder atonia, neurogenic bladder disorder or other neurological disorder that is impacting bladder function (eg multiple sclerosis, Parkinson's disease, spinal cord injuries, etc)
* Urethral stricture, bladder neck contracture, sphincter abnormalities, urinary obstruction due to causes other than BPH, or other potentially confounding bladder or urethral disease or condition
* Allergy to iodinated contrast agents
* Hypersensitivity to gelatin products
* Previous non-medical BPH treatment, including surgery, TURP, needle ablation, microwave or laser therapy, balloon dilation, stent implantation, or any other invasive treatment to the prostate
* Known major iliac arterial occlusive disease or any known condition that catheterization of the prostatic arteries or is a contraindication to embolization, as vasospasm, anatomical variations that imply a risk of embolization, bleeding, prostatic arteries diameter inferior to microcatheter profile, pelvic inflammatory disease
* Contraindication to magnetic resonance imaging
* History of prostatitis in the last 5 years, not totally controlled with medical treatment
* History of pelvic irradiation or radical pelvic surgery
* Coagulation disturbances not normalized by medical treatment

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms | 12 months
  Improvement (change) of symptoms assessed by IPSS Score (International Prostate Symptom Score )

SECONDARY OUTCOMES:
Improvement in QoL | 12 months
  Improvement (change) of quality of life assessed by QoL score
Duration of hospitalization post procedure | 3 weeks
  Number of days of postprocedure hospitalization
Preservation of erectile function | 12 months
  Change from baseline in erectile function using the International Index of Erectile Function (IIEF)

OTHER OUTCOMES:
Maximum urinary flow rate | 12 months
  Change from baseline in maximum urinary flow rate (Qmax)
Post-void residual urinary volume | 12 months
  Change from baseline in post-void residual urinary volume (PVR)
Detrusor pressure | 12 months
  Change from baseline in detrusor pressure (Pdet)
Mean prostate volume | 12 months
  Change from baseline in mean prostate volume, as determined by transrectal US
Structural and morphological changes in MRI | 12 months
  Change from baseline in mean prostate volume, and structural and morphological changes as determined by MRI
Prostate specific antigen | 12 months
  Change from baseline in prostate specific antigen (PSA)
Overall adverse events | 12 months
  Overall adverse events
Procedure related adverse events | 12 months
  Procedure related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A De Gregorio, PhD, Principal Investigator — University of Zaragoza. Chairman of Radiology
Locations (1):
- Hospital Universitario Lozano Blesa, Zaragoza, Spain